CLINICAL TRIAL: NCT07105761
Title: Effects of Body-mind-spirit Group Therapy on Holistic Well-being and Depression in Individuals With Visual Impairment
Brief Title: Body-Mind-Spirit Action Group on the Well-being
Acronym: BMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chuen-Ru Liu, Registered Nurse in Public Service, Taipei City Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: TCHIRB-11107010
Record Dates: First submitted 2025-07-18; First posted 2025-08-06 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Quality of Life (QOL); Depression
Keywords: Body-mind-spirit; group therapy; quality of life; sleep quality; depression; holistic well-being
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study employed a quasi-experimental design with matched groups, where participants were assigned to either the intervention or the control group based on their registration order and availability
Masking Description: Measurement points were set at weeks 1, 5, and 10 during the intervention. The study was approved by the Institutional Review Board of Taipei City Hospital Research Ethics Committee (Taiwan) (TCHIRB-11107010) and adheres to the ethical guidelines of the Declaration of Helsinki.This study employed a quasi-experimental design with matched groups, where participants were assigned to either the intervention or the control group based on their registration order and availability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body-Mind-Spirit (Experimental): The experimental group participated in a 10-week BMS group intervention , consisting of weekly 130-minute sessions that incorporated thematic discussions, mindfulness practices, therapeutic storytelling, and gratitude/forgiveness activities tailored to the needs of individuals with visual impairment.
  Interventions: Behavioral: Body-Mind-Spirit
- routine activities (No Intervention): Ｔhe control group participated in routine activities without body-mind-spirit intervention

INTERVENTIONS:
Behavioral: Body-Mind-Spirit — The experimental group participated in a 10-week BMS group intervention, with weekly 130-minute sessions. The intervention combined Eastern philosophy and Western psychotherapy to enhance emotional balance and psychological resilience. Core components included observing merits (recognizing strengths), cultivating gratitude, and practicing forgiveness. Physical activities such as finger dexterity training, diaphragmatic breathing, and stretching supported autonomic regulation and flexibility. Psychological strategies involved positive thinking, emotional expression, and life story sharing. All materials were adapted with audio descriptions for accessibility. Participants with visual impairment received orientation training and volunteer support for transportation and on-site assistance.
  Arms: Body-Mind-Spirit

SUMMARY:
Primary Purpose:

To evaluate the effectiveness of a culturally adapted BMS group intervention on holistic well-being, depressive symptoms, sleep parameters, and quality of life in individuals with visual impairment.

Study Objective:

This study aims to find out whether a 10-week BMS group program can help people with visual impairment feel emotionally better, improve their overall well-being, enhance sleep quality, and experience a higher quality of life.

Intervention Description:

The BMS group meets once a week for 10 weeks, with each session lasting about 2 hours. Sessions include guided discussions, storytelling, and experiential activities drawn from both Eastern and Western philosophies. These practices focus on:

Appreciating kindness in others Letting go of past hurt (forgiveness) Practicing mindfulness and living in the present moment

What the Researchers Want to Know:

Does the program help participants feel less depressed? Does it help them feel more balanced, hopeful, and connected in daily life? Does it improve their sleep and overall well-being?

Participants:

About 30 community-dwelling adults with visual impairment will take part in the study. They will be randomly assigned to one of two groups:

The intervention group will join the BMS sessions for 10 weeks. The control group will continue their usual community activities with no new program.

All participants will complete surveys at three points: before the program starts, at the midpoint (week 5), and after the program ends (week 10). These surveys assess levels of depression, well-being, sleep quality, and life satisfaction. Some participants in the BMS group will also be invited to join short interviews to share their experiences-such as feeling more grateful, confident, or resilient.

Overall Goal:

The goal of this study is to determine whether a supportive, culturally adapted group program can help people with vision loss feel stronger, less depressed, more connected, and better equipped to manage their daily lives. Previous findings suggest that BMS group therapy effectively enhances sleep duration and significantly improves quality of life-especially in psychological well-being-among visually impaired individuals. These findings support the integration of BMS therapy into holistic care strategies to promote emotional resilience, well-being, and personal growth in this population.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a culturally adapted BMS group intervention on holistic well-being, depressive symptoms, sleep quality, and overall quality of life among individuals with visual impairment. The BMS model integrates principles of Eastern and Western psychological and spiritual care. Through practices such as awareness cultivation, forgiveness, gratitude, and mindfulness, it seeks to enhance emotional resilience and psychological recovery.

A quasi-experimental controlled design will be adopted. Thirty community-dwelling adults with visual impairment will be recruited and randomly assigned to either an intervention group or a control group. The intervention group will participate in a 10-week BMS group program, meeting once a week for approximately two hours per session. Each session includes thematic discussions, mindfulness exercises, therapeutic storytelling, and activities focused on gratitude and forgiveness. All materials and course designs are adapted to meet the specific needs of individuals with visual impairment and are delivered by a trained professional team.

All participants will complete standardized questionnaires at three time points: pre-intervention (baseline), mid-intervention (week 5), and post-intervention (week 10). These assessments will measure levels of depression, psychological well-being, sleep quality, and life satisfaction. In addition, a subset of participants from the intervention group will be invited to participate in interviews to collect qualitative data and supplement quantitative findings.

This study aims to explore the potential mechanisms by which BMS intervention promotes psychological health and quality of life in individuals with visual impairment. The findings may serve as empirical support for the development of non-pharmacological mental health interventions and community care models, offering valuable implications for practice and policy advancement.

ELIGIBILITY:
Inclusion Criteria:

1. Possession of a valid disability certificate indicating visual impairment
2. Age between 20 and 95 years
3. Provision of informed consent by both the participant and their legal guardian
4. Willingness to participate in group discussions and to consent to the audio recording of sessions
5. Ability to communicate verbally

Exclusion Criteria:

1. Presence of deafness or muteness that prevents effective verbal communication
2. Current involvement in any form of psychological or group therapy
3. A Mini-Mental State Examination (MMSE) score below 3, indicating an inability to express personal intentions verbally.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Holistic Well-being Scale (HWS) | Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 10)
  The HWS scale comprises 30 items designed to assess the physical, psychological, and spiritual dimensions that enhance life satisfaction and well-being. It evaluates two major constructs:
  1. Perceived affliction, including psychological vulnerability, bodily irritability, and spiritual disorientation
  2. Equanimity, including vitality, mindful awareness, non-attachment, and spiritual self-care Participants respond on a scale from 0 (complete disagreement) to 10 (complete agreement) for each item. Higher scores on perceived affliction indicate lower spiritual resilience, while higher scores on equanimity indicate greater spiritual resilience and well-being.
Beck Depression Inventory-II scores(BDI-II) | Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 10)
  The BDI-II scores is a self-administered 21-item questionnaire designed to assess the severity of depressive symptoms. Each item is scored on a scale from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms (worse outcome)
World Health Organization Quality of Life Questionnaire-Taiwan version (WHOQOL-BREF TW) | Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 10)
  The WHOQOL-BREF TW is a 28-item questionnaire assessing four domains: physical health (7 items), psychological well-being (6 items), social relationships (4 items), and environmental factors (9 items). Each item uses a 5-point Likert scale, with higher scores indicating better quality of life. Domain scores are calculated by summing the item scores within each domain, multiplying by 4, and dividing by the number of items, resulting in scores ranging from 4 to 20. Higher scores represent better quality of life. This questionnaire provides a comprehensive reflection of an individual's multidimensional health status and subjective satisfaction, making it suitable for people with visual impairments..
sleep quality | Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 10)
  Subjective Assessment of Sleep Quality To evaluate participants' perceived sleep quality, this study utilized Item 16 from the WHOQOL-BREF Taiwan version, which asks: "Are you satisfied with your sleep?" Responses were rated on a 5-point Likert scale, reflecting overall subjective satisfaction with sleep Objective Assessment of Sleep Quality Objective sleep parameters were measured using a wrist-worn accelerometer (e.g., XA-5), which recorded data on total sleep time, sleep efficiency, and nighttime awakenings. The device estimates sleep states based on three-axis movement patterns.
qualitative inquiry | Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 10)
  The question design was informed by Yalom's recommendations regarding therapeutic mechanisms and primarily addressed the following topics: participants' personal definitions of well-being; whether well-being improved after attending the program and in which specific dimensions (physical, mental, and spiritual); experience of growth and transformation before and after participation; the most impressive and interesting event that occurred in the group; and suggestions for enhancing the practicality and adaptability of the course content

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Ru Liu, PhD, Study Chair — Taipei City Hospital Songde Branch
Locations (1):
- Chinese Visually Impaired Anyang Welfare Association, Taipei, No. 37, Yining St., Datong Dist.,, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
1. Quantitative Data
     Pre- and Post-Measurement Scores:
     Tool A: Pre-test, Post-test Tool B: Pre-test, Post-test Tool C: Pre-test, Post-test
  2. Attendance Rate and Participation Records Attendance Rate: Percentage of participants attending each intervention session.
     Participation Records: Number of participation sessions and times for each participant.
  3. Data Availability Timeline and Conditions Availability Timeline: Applications will open 6 months after the main results are published.
     Usage Conditions:
     Data is available only to researchers approved by IRB or ethical review. Research purposes must be clear and comply with ethical standards.
  4. Research Results Summary of Results: Analyze the impact of changes in pre- and post-test scores on participants.
  Statistical Analysis: Use t-tests or ANOVA to assess group differences. Qualitative Analysis: Conduct thematic analysis on participant feedback
Supporting Information: Study Protocol, CSR
Time Frame: July 2025 - July 2026
Access Criteria: Who can access the data:
  Qualified researchers affiliated with academic institutions or research organizations may request access to the individual participant data and supporting documents.
  What information they can access:
  De-identified individual participant data related to the outcomes reported in this study, including supporting documents such as the study protocol, statistical analysis plan, informed consent form, and data dictionary.
  How they can access the data:
  Interested researchers must submit a formal data access request including a research proposal, data use plan, and documentation of ethics approval. Upon review and approval by the data access committee, data will be made available through a secure data-sharing platform under a data use agreement.
URL: https://zenodo.org/records/15862065

REFERENCES:
- [Background] Yeh HC, Yang S, Fu JS, et al. Developing college students' critical thinking through reflective writing. Higher Educ Res Dev. 2023;42(1):244-259. doi: 10.1080/07294360.2022.2043247.
- [Background] Martínez-Martí ML, Hernández-Lloreda MJ, Avia MD. Appreciation of beauty and excellence: relationship with personality, prosociality, and well-being. J Happiness Stud. 2016;17(6):2613-2634. doi: 10.1007/s10902-015-9709-6.
- [Background] Ho CYY, Yu BCL, Mak WWS. Nonattachment mediates the associations between mindfulness, well-being, and psychological distress: A meta-analytic structural equation modeling approach. Clin Psychol Rev. 2022 Jul;95:102175. doi: 10.1016/j.cpr.2022.102175. Epub 2022 Jun 3. PMID 35690041
- [Background] Zamzam AM. Understanding the correlation between visual impairment and mental health: a literature review. Sriwijaya J Ophthalmol. 2021;4(1):58-63. doi: 10.37275/sjo.v4i1.57.
- [Background] Martina BI, Mazzi C, Colombari E, et al. The interplay between visual perception and psychopathological conditions in adult patients: a systematic review. J Psychosom Res. 2024;181:111709.
- [Background] Demmin DL, Silverstein SM. Visual Impairment and Mental Health: Unmet Needs and Treatment Options. Clin Ophthalmol. 2020 Dec 3;14:4229-4251. doi: 10.2147/OPTH.S258783. eCollection 2020. PMID 33299297
- See also: Storage of study design, informed consent forms, study rota, and study results. — https://zenodo.org/records/15862065
- Available data/document: Study Protocol: 15862065 — https://zenodo.org/records/15862065 — The de-identified individual participant data (IPD) and supporting documents will be available to qualified researchers upon request, following review and approval by a data access committee. Data will be shared via a secure institutional repository beginning 6 months after study completion, for up to 3 years.